CLINICAL TRIAL: NCT04299425
Title: Evaluating Impact of Near Infrared Autofluorescence (NIRAF) Detection for Identifying Parathyroid Glands During Parathyroidectomy
Brief Title: Evaluating Impact of NIRAF Detection for Identifying Parathyroid Glands During Parathyroidectomy
Acronym: NIRAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Carmen Solorzano, Professor of Surgery Chair, Department of Surgery Director, Vanderbilt Endocrine Surgery, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB 192486; 5R01CA212147-02 (NIH)
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Results first posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-04

CONDITIONS: Parathyroid Adenoma; Parathyroid Neoplasms; Parathyroid Hyperplasia; Parathyroid Cancer; Hypercalcemia; Primary Hyperparathyroidism
Keywords: Parathyroidectomy; Intraoperative Parathyroid Identification; Near Infrared Autofluorescence; Persistent Hyperparathyroidism; Persistent Hypercalcemia; Failed Parathyroidectomy; Repeat Parathyroidectomy
MeSH Terms: conditions — Parathyroid Neoplasms; Hypercalcemia; Hyperparathyroidism, Primary

STUDY DESIGN:
Intervention Model Description: NIRAF detection technology is used as an adjunctive tool for intraoperative parathyroid identification in patients who undergo parathyroidectomy (PTx) in the interventional group.
  Generic Name of Device: Parathyroid Autofluorescence Detection Device (NIRAF detection technology).
  The Parathyroid Autofluorescence Detection Device consists of a disposable fiber-optic probe that emits non-ionizing radiation from a near infrared (NIR) 785 nanometer (nm) laser source, and also transmits the resulting tissue NIRAF to a photo-detector. The 785 nm laser source emits a maximum power of 20 milliwatts (mW). The device has an FDA clearance for clinical use in general surgeries and dermatological use (Class 2 device).
Who Masked: Participant
Masking Description: Only participants will be masked to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- NIRAF Detection Technology + (Experimental): Parathyroid gland identification will be performed with PTeye using NIRAF detection technology as an adjunctive tool in patients who undergo parathyroidectomy (PTx).
  Interventions: Device: NIRAF Detection Technology
- NIRAF Detection Technology - (No Intervention): Parathyroid gland identification will be performed with the naked eye of the surgeon without using PTeye - NIRAF detection technology in patients who undergo parathyroidectomy (PTx).

INTERVENTIONS:
Device: NIRAF Detection Technology — Near Infrared Autofluorescence (NIRAF) detection technology or 'PTeye' consists of a disposable fiber-optic probe that emits non-ionizing radiation from a NIR 785 nm laser source, and also transmits the resulting tissue NIRAF to a photo detector. The 785 nm laser source emits a maximum power of 20 mW. The device is FDA cleared for clinical use in general surgeries and dermatological use (Class 2 device).
  After surgeon identifies a potential parathyroid gland in the surgical field, the surgeon places the fiber-optic probe of PTeye on suspect tissue and presses the device foot-pedal to activate tissue NIRAF measurement. Auditory beep at high frequency with a Detection Ratio > 1.2 is interpreted by device as the suspect tissue being positive for parathyroid.
  Other Names: PTeye Device
  Arms: NIRAF Detection Technology +

SUMMARY:
This study describes a single center, randomized, single-blinded clinical trial to assess the clinical benefits of the use of near infrared autofluorescence (NIRAF) detection with an FDA-cleared device 'Parathyroid Eye (PTeye)' for identifying parathyroid glands (PGs) during parathyroidectomy (PTx) procedures. It compares risk-benefits and outcomes in PTx patients where NIRAF detection with PTeye for parathyroid identification is either used or not used.

DETAILED DESCRIPTION:
Inability of the surgeon to identify or localize the diseased PG can occur in 5 - 10% of cases resulting in failed parathyroidectomies (PTx). As a result, persistent hyperparathyroidism can occur in these patients resulting in unnecessary repeat surgeries that may be associated with increased morbidity and costs. Ultrasound imaging, 99mTechnetium-sestamibi scintigraphy, and computed tomography (CT) have so far demonstrated variable efficacy in preoperative localization of diseased PGs and may not always correlate well with the surgical field of view as observed intraoperatively. Consequently, most surgeons rely on visual identification of PGs during surgery, whereby the accuracy of PG identification is eventually determined by her/his surgical skill and experience. When in doubt, a surgeon routinely confirms the identity of PG tissue intraoperatively by sending the specimen for frozen section analysis that typically requires a wait time of 20-30 minutes per sample and has additional costs.

By easily being able to distinguish parathyroid from other tissues intraoperatively, postsurgical complications and associated costs may be reduced. The unique discovery of near infrared autofluorescence (NIRAF) in parathyroid tissues demonstrated that optical modalities that detect NIRAF can be utilized for non-invasive and label-free identification of parathyroid tissues with an accuracy as high as 97%. Since then, several research groups have explored the feasibility of localizing parathyroid glands using NIRAF detection with reasonable success, resulting in FDA clearance for marketing this optical technique. In this study, we plan to evaluate whether an FDA-cleared device called 'PTeye' (AiBiomed, Santa Barbara, CA) is beneficial or not, for the surgeon and patient during PTx operations. The results of such a study will help us to understand and assess the true impact of optical modalities such as PTeye on (i) improving the quality and efficiency of PTx surgeries and (ii) minimizing risk of postsurgical complications and related expenses.

The aim of this prospective single blinded randomized study is to compare 2 groups of patients: PTx patients operated using NIRAF detection technology with PTeye as adjunct tool (NIRAF+) vs. patients operated without the adjunct technology (NIRAF-). The main objective of this study is to assess the benefit of intraoperative use of NIRAF detection technology via PTeye during PTx procedures with regard to PG identification, duration of surgery, number of frozen section analysis performed, number of intraoperative PTH assays sent and incidence of postsurgical complications, if any and history of ER visits or hospitalization or repeat surgeries due to persistent high blood calcium after PTx procedure, compared to standard of care.

ELIGIBILITY:
Inclusion Criteria:

* All primary hyperparathyroidism patients eligible for parathyroidectomy (PTx). Both bilateral and focused mode of PTx will be considered for this study, based on the surgeon's preference.
* Re-operative primary hyperparathyroidism patients who have undergone a failed prior PTx.

Exclusion Criteria:

* Patients with concurrent parathyroid and thyroid disease that require total thyroidectomy.
* Patients with secondary or tertiary hyperparathyroidism.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen C Solorzano, MD, FACS, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Informed Consent Form and Clinical Study Report will be made available to other researchers as per the specified time-frame
Supporting Information: ICF, CSR
Time Frame: Clinical Study Report will be shared 6 months after publication of trial data and will be available till end date of trial. Informed Consent Form will be shared for a year after the primary completion date of the trial.
Access Criteria: Request for Individual Patient Data (IPD) - Informed consent Form and Clinical Study Report - will be reviewed by the principal investigator of this clinical trial, before granting access to IPD

REFERENCES:
- [Background] Simental A, Ferris RL. Reoperative parathyroidectomy. Otolaryngol Clin North Am. 2008 Dec;41(6):1269-74, xii. doi: 10.1016/j.otc.2008.05.008. PMID 19040985
- [Background] Cron DC, Kapeles SR, Andraska EA, Kwon ST, Kirk PS, McNeish BL, Lee CS, Hughes DT. Predictors of operative failure in parathyroidectomy for primary hyperparathyroidism. Am J Surg. 2017 Sep;214(3):509-514. doi: 10.1016/j.amjsurg.2017.01.012. Epub 2017 Jan 10. PMID 28108069
- [Background] Doherty GM, Weber B, Norton JA. Cost of unsuccessful surgery for primary hyperparathyroidism. Surgery. 1994 Dec;116(6):954-7; discussion 957-8. PMID 7985102
- [Background] Wachtel H, Cerullo I, Bartlett EK, Kelz RR, Karakousis GC, Fraker DL. What Can We Learn from Intraoperative Parathyroid Hormone Levels that Do Not Drop Appropriately? Ann Surg Oncol. 2015;22(6):1781-8. doi: 10.1245/s10434-014-4201-9. Epub 2014 Oct 30. PMID 25354574
- [Background] Mohebati A, Shaha AR. Imaging techniques in parathyroid surgery for primary hyperparathyroidism. Am J Otolaryngol. 2012 Jul-Aug;33(4):457-68. doi: 10.1016/j.amjoto.2011.10.010. Epub 2011 Dec 7. PMID 22154018
- [Background] Ahuja AT, Wong KT, Ching AS, Fung MK, Lau JY, Yuen EH, King AD. Imaging for primary hyperparathyroidism--what beginners should know. Clin Radiol. 2004 Nov;59(11):967-76. doi: 10.1016/j.crad.2004.04.005. PMID 15488844
- [Background] Sosa JA, Powe NR, Levine MA, Udelsman R, Zeiger MA. Profile of a clinical practice: Thresholds for surgery and surgical outcomes for patients with primary hyperparathyroidism: a national survey of endocrine surgeons. J Clin Endocrinol Metab. 1998 Aug;83(8):2658-65. doi: 10.1210/jcem.83.8.5006. PMID 9709928
- [Background] Chen H, Wang TS, Yen TW, Doffek K, Krzywda E, Schaefer S, Sippel RS, Wilson SD. Operative failures after parathyroidectomy for hyperparathyroidism: the influence of surgical volume. Ann Surg. 2010 Oct;252(4):691-5. doi: 10.1097/SLA.0b013e3181f698df. PMID 20881776
- [Background] Novis DA, Zarbo RJ. Interinstitutional comparison of frozen section turnaround time. A College of American Pathologists Q-Probes study of 32868 frozen sections in 700 hospitals. Arch Pathol Lab Med. 1997 Jun;121(6):559-67. PMID 9199619
- [Background] McWade MA, Sanders ME, Broome JT, Solorzano CC, Mahadevan-Jansen A. Establishing the clinical utility of autofluorescence spectroscopy for parathyroid detection. Surgery. 2016 Jan;159(1):193-202. doi: 10.1016/j.surg.2015.06.047. Epub 2015 Oct 9. PMID 26454675
- [Background] McWade MA, Paras C, White LM, Phay JE, Mahadevan-Jansen A, Broome JT. A novel optical approach to intraoperative detection of parathyroid glands. Surgery. 2013 Dec;154(6):1371-7; discussion 1377. doi: 10.1016/j.surg.2013.06.046. PMID 24238054
- [Background] Voelker R. Devices Help Surgeons See Parathyroid Tissue. JAMA. 2018 Dec 4;320(21):2193. doi: 10.1001/jama.2018.18768. No abstract available. PMID 30512085
- [Derived] Cousart AG, Kiernan CM, Willmon PA, Thomas G, Wang TS, Gauger PG, Duh QY, Underwood HJ, Jackson A, Patel A, Mahadevan-Jansen A, Solorzano CC. Near-Infrared Autofluorescence for Parathyroid Detection During Endocrine Neck Surgery: A Randomized Clinical Trial. JAMA Surg. 2025 Sep 1;160(9):936-944. doi: 10.1001/jamasurg.2025.2233. PMID 40668552

RESULTS

PARTICIPANT FLOW:
Groups:
- NIRAF Detection Technology +: Parathyroid gland identification will be performed with PTeye using NIRAF detection technology as an adjunctive tool in patients who undergo parathyroidectomy (PTx).
  NIRAF Detection Technology: Near Infrared Autofluorescence (NIRAF) detection technology or 'PTeye' consists of a disposable fiber-optic probe that emits non-ionizing radiation from a NIR 785 nm laser source, and also transmits the resulting tissue NIRAF to a photo detector. The 785 nm laser source emits a maximum power of 20 mW. The device is FDA cleared for clinical use in general surgeries and dermatological use (Class 2 device).
  After surgeon identifies a potential parathyroid gland in the surgical field, the surgeon places the fiber-optic probe of PTeye on suspect tissue and presses the device foot-pedal to activate tissue NIRAF measurement. Auditory beep at high frequency with a Detection Ratio > 1.2 is interpreted by device as the suspect tissue being positive for parathyroid.
Period: Overall Study
Arm/Group | NIRAF Detection Technology + | NIRAF Detection Technology -
Started | 80 | 80
Completed | 80 | 80
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NIRAF Detection Technology + | NIRAF Detection Technology - | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (14.6) | 59.8 (14.4) | 58.3 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 63 | 125
  Male | 18 | 17 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 73 | 74 | 147
  Black | 5 | 6 | 11
  Asian | 1 | 0 | 1
  Other | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic | 79 | 80 | 159
  Hispanic | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 80 | 80 | 160
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 30.77 (7.52) | 30.94 (7.72) | 30.85 (7.59)
Diagnosis [Count of Participants; unit: Participants]
  Primary sporadic HPT | 72 | 71 | 143
  Persistent HPT | 3 | 9 | 12
  Recurrent HPT | 1 | 0 | 1
  MEN1 | 2 | 0 | 2
  Parathyroid carcinoma | 1 | 0 | 1
  Lithium-induced HPT | 1 | 0 | 1
Preoperative calcium (pg/dL) [Mean (Standard Deviation); unit: mg/dL] | 11.115 (0.689) | 11.112 (0.712) | 11.112 (0.712)
Preoperative PTH (pg/mL) [Mean (Standard Deviation); unit: pg/mL] | 152.3 (79.8) | 163.6 (139) | 157.9 (112.7)
Preoperative vitamin D [Mean (Standard Deviation); unit: mcg] | 36.7 (16) | 39.6 (20.5) | 38.1 (18.2)
Procedure by intention [Count of Participants; unit: Participants]
  Focused | 27 | 24 | 51
  Bilateral | 53 | 56 | 109

OUTCOME MEASURES:

1. Primary Outcome: Average Number of Parathyroid Glands Identified With High Confidence Per Patient
Description: Average number of parathyroid glands identified (Experimental Group: Glands identified with naked eye + NIRAF; Control Group: Glands identified with naked eye) per patient
Time Frame: Immediate. During PTx procedure.
Measure: Mean (Standard Deviation); unit: parathyroid glands
Arm/Group | NIRAF Detection Technology + | NIRAF Detection Technology -
Number analyzed (Participants) | 80 | 80
parathyroid glands | 3.1 (1.21) | 2.7 (1.13)
Statistical Analysis 1: Comparison: NIRAF Detection Technology + vs NIRAF Detection Technology -; Test type: Superiority; p = 0.04, t-test, 2 sided

2. Secondary Outcome: Number of Participants With Persistent Hyperparathyroidism or Hypercalcemia (Failed Parathyroidectomy).
Description: If blood calcium with/without parathyroid hormone (PTH) has not normalized at 1st post-operative visit, calcium and/or PTH is subsequently measured as necessary. Patient is defined to have a failed parathyroidectomy if hypercalcemia/hyperparathyroidism (defined as total blood calcium level > 10.5 mg/dL or 2.6 mmol/L, with/without elevated serum intact PTH > 65 pg/ml or 6.9 pmol/L) persists at or after the 6th postoperative month.
Time Frame: 6 months after PTx procedure
Measure: Count of Participants; unit: Participants
Arm/Group | NIRAF Detection Technology + | NIRAF Detection Technology -
Number analyzed (Participants) | 80 | 80
Participants | 0 | 1
Statistical Analysis 1: Comparison: NIRAF Detection Technology + vs NIRAF Detection Technology -; Test type: Superiority; p = 1.0, Chi-squared

3. Secondary Outcome: Number of Frozen Sections Sent for Analysis
Description: Number of frozen sections sent for analysis during the procedure to confirm potential parathyroid tissue
Time Frame: Immediate. During PTx procedure.
Measure: Number; unit: frozen sections
Arm/Group | NIRAF Detection Technology + | NIRAF Detection Technology -
Number analyzed (Participants) | 80 | 80
frozen sections | 13 | 45

4. Secondary Outcome: Duration of Parathyroidectomy (PTx) Procedure
Description: Duration of PTx procedure - timed from skin incision until the surgeon notifies the anesthesia team to awaken the patient
Time Frame: Immediate. During PTx procedure.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | NIRAF Detection Technology + | NIRAF Detection Technology -
Number analyzed (Participants) | 80 | 80
minutes | 89.3 (32.6) | 95.5 (39.7)
Statistical Analysis 1: Comparison: NIRAF Detection Technology + vs NIRAF Detection Technology -; Test type: Superiority; p = 0.55, t-test, 2 sided

5. Secondary Outcome: Number of Participants Stratified by Duration of Hospital Stay
Description: Number of nights spent for postoperative recovery in the hospital after the surgical procedure.
Time Frame: 0-72 hours after PTx procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | NIRAF Detection Technology + | NIRAF Detection Technology -
Number analyzed (Participants) | 80 | 80
Participants
  Discharged same day | 64 | 66
  Overnight | 14 | 14
  Admitted > 23 hours | 2 | 0
Statistical Analysis 1: Comparison: NIRAF Detection Technology + vs NIRAF Detection Technology -; Test type: Superiority; p = 0.36, Chi-squared

6. Secondary Outcome: Number of 'False Positive' Tissues Excised by Surgeon
Description: Number of tissues that were excised by surgeon assumed to be parathyroid tissue, but is later validated as non-parathyroid tissue (false positive) by histology
Time Frame: Immediate to 10 days after PTx procedure.
Population: Only the NIRAF Detection Technology + arm was included in the analysis to calculate the rate of false positives by the device. Since the NIRAF Detection Technology - did not use the device that arm was not included.
Measure: Number; unit: false positives
Arm/Group | NIRAF Detection Technology +
Number analyzed (Participants) | 80
false positives | 19

7. Secondary Outcome: Number of Patients Who Have Had Repeat Parathyroidectomy (PTx) Procedure
Description: Number of patients with repeat PTx procedure performed after the current procedure.
Time Frame: At 6-months post-operation
Population: Nearly all patients attended their first follow-up appointment (5-14 days post-operation), however about 30 patients were lost for long-term follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | NIRAF Detection Technology + | NIRAF Detection Technology -
Number analyzed (Participants) | 51 | 50
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 2 years, 5 months.
Arm/Group | NIRAF Detection Technology + | NIRAF Detection Technology -
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 0/80 | 0/80

LIMITATIONS AND CAVEATS:
Only 63% of the cohort had follow-up for 6-months or longer, which may underestimate the rate of failure. The relatively small sample size may miss rare events such as operative failure. Additionally, inter-variability amongst the two surgeons and their surgical approaches adds more complexity. Lastly, these findings may only be generalizable to higher volume centers with more experienced surgeons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/25/NCT04299425/Prot_SAP_002.pdf
  • Informed Consent Form (2021-01-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT04299425/ICF_001.pdf